CLINICAL TRIAL: NCT00814372
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Study to Evaluate the Safety and Efficacy of MBX-102/JNJ-39659100 in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: Evaluate Safety and Effectiveness of MBX-102 in Type 2 Diabetes Patients With Poor Glycemic Control on Metformin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: MBX-102 did not meet the target efficacy profile of HbA1c change.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M102-20814
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — arhalofenate; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MBX-102 400 (Experimental)
  Interventions: Drug: MBX-102; Drug: Metformin
- MBX-102 600 (Experimental)
  Interventions: Drug: MBX-102; Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Metformin
- Actos (Active Comparator): 30-45 mg
  Interventions: Drug: Actos; Drug: Metformin

INTERVENTIONS:
Drug: MBX-102 — capsule
  Arms: MBX-102 400; MBX-102 600
Drug: Placebo — matching placebo
  Arms: Placebo
Drug: Actos — over-encapsulated to match MBX-102 and placebo
  Arms: Actos
Drug: Metformin — greater than or equal to 1500 mg/kg day

SUMMARY:
To define the relative efficacy, safety and tolerability profiles of oral daily MBX-102 at daily doses of 400 and 600 mg vs. placebo and Actos® 30 mg (up-titrated to 45 mg after 8 weeks) when administered for up to 24 weeks in patients inadequately controlled with a stable dose of metformin (≥ 1500 mg/day).

DETAILED DESCRIPTION:
Approximately 240 patients will be randomized in this study, 60 to each of two MBX-102 treatment groups (400 and 600 mg daily), 60 to placebo, and 60 to the Actos® group. Patients in the Actos® group will receive Actos® 30 mg/daily for the first eight weeks of the treatment phase and Actos® 45 mg/daily for the last 16 weeks of the treatment phase. Patients in the MBX-102 400 mg group and MBX-102 600 mg group will continue MBX-102 400 mg and 600 mg, respectively for the full 24 weeks. All study medication will be over-encapsulated; thus, each patient will take two blinded capsules each day containing either placebo, MBX-102 or Actos®. This sample size provides the minimum number expected to ensure a power of at least 90% in detecting a difference of 0.64% in HbA1c between the placebo and experimental treatment, using a two-tailed, two-sample t-test with type 1 error of 0.05, when the pooled standard deviation is ≤ 1.0%, and the discontinuation rate is ≤ 12.5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who have been on metformin for the last 6 months and are taking a stable dose of metformin (≥ 1500 mg/d) as monotherapy for at least the last 3 months
* Male or female, 18-70 years of age
* All female patients must be surgically sterile or post-menopausal (at least 40 years of age with no history of menses for at least 2 years; or any age with no history of menses for at least 6 months and serum FSH ≥ 40 mIU/mL) or must agree to use two medically accepted methods of contraception including a barrier method. Depo contraceptives are excluded.
* Female patients must not be pregnant or lactating
* BMI ≥ 26 (patients of Asian Indian origin ≥ 22) kg/m2
* HbA1c ≥ 7.5%, ≤ 10.5%
* FPG ≥ 120 mg/dL, ≤ 240 mg/dL

Exclusion Criteria:

* History of diabetes secondary to pancreatitis or pancreatectomy
* Any history of ketoacidosis
* History of insulin use within last one year (insulin use while hospitalized is acceptable)
* Weight loss > 10 pounds in the three months prior to screening visit
* History of TZD use (Actos® or Avandia®) within 6 months of screening visit
* History of TZD discontinuation due to side effect or lack of efficacy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline and compared to placebo | 24 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG) from baseline and vs. placebo | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Denham, M.D., Principal Investigator — dgd Research, Inc.; Thomas W. Littlejohn, M.D., Principal Investigator — Piedmont Medical Research Associates; Michael Guice, M.D., Principal Investigator — American Institute of Research; K. M. Prasanna Kumar, MD, Principal Investigator — M. S. Ramaiah Memorial Hospital; Veerasamy Seshiah, MD, Principal Investigator — Dr. V. Seshiah Diabetes Care & Research Institute; Sanjay Kalra, MD, Principal Investigator — Bharti Research Institute of Diabetes & Endocrinology; Sailesh Lodha, MD, Principal Investigator — Fortis Hospital; Ariachery C Ammini, MD, Principal Investigator — All India Institute of Medical Sciences; Prema Varthakavi, MD, Principal Investigator — BYL Nair Hospital; Sanjiv Shah, MD, Principal Investigator — Diabetes Action Centre; Manoj Chadha, MD, Principal Investigator — PD Hindhuja National Hospital & Medical Research Centre; Mathew Thomas, MD, Principal Investigator — Health & Research Centre; Sanjay Reddy, MD, Principal Investigator — Bangalore Diabetes Centre; Ganapati Bantwal, MD, Principal Investigator — St Johns Medical College Hospital, Bangalore, India; Aravind S Sosale, MD, Principal Investigator — Diacon Hospital Diabetes & Research Centre; Vaishali Deshmukh, MD, Principal Investigator — Deenanath Mangeshkar Hospital & Research Centre; Abhay Mutha, MD, Principal Investigator — Diabetes Care & Research Centre; Nihal Thomas, MD, Principal Investigator — Christian Medical College, Vellore, India; Kirtikumar Modi, MD, Principal Investigator — Medwin Hospital; Sunil Jain, MD, Principal Investigator — Diabetes Thyroid Hormone Research Institute Pvt. Ltd.; Pramod Gandhi, MD, Principal Investigator — Gandhi Endocrinology & Diabetes Centre; Rakesh Kumar Sahay, MD, Principal Investigator — Mediciti Hospital; Harish Kumar, MD, Principal Investigator — Amrita Institute of Medical Sciences; Rubin Savedra, MD, Principal Investigator — Association of International Professionals, dba Nevada Alliance Against Diabetes; Teresa Sligh, MD, Principal Investigator — Translational Research Group, Inc. dba Providence Clinical Research; Prabha Adhikari, MD, Principal Investigator — Kasturba Medical College Hospital; Navneet Agrawal, MD, Principal Investigator — Diabetes, Obesity and Thyroid Center; Swamy Miryala, MD, Principal Investigator — Kamineni Hospitals Pvt, Ltd.
Locations (26):
- United States (5):
  - Providence Clinical Research, Burbank, California
  - American Institute of Research, Los Angeles, California
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - DGD Research, Inc., San Antonio, Texas
- India (21):
  - Kamineni Hospitals Pvt, Ltd., Hyderabad, Andhra Pradesh
  - Bangalore Diabetes Centre, Bangalore
  - Diacon Hospital Diabetes & Research Centre, Bangalore
  - M. S. Ramaiah Memorial Hospital, Bangalore
  - St. John's Medical College & Hospital, Bangalore
  - Dr. V. Seshiah Diabetes Care & Research Institute, Chennai
  - Mediciti Hospital, Hyderabad
  - Medwin Hospital, Hyderabad
  - Diabetes Thyroid Hormone Research Institute Pvt. Ltd., Indore
  - Fortis Hospital, Jaipur
  - Bharti Research Institute of Diabetes & Endocrinology, Karnāl
  - Amrita Institute of Medical Sciences, Kochi
  - Diabetes Action Centre, Mumbai
  - BYL Nair Hospital, Mumbai
  - PD Hindhuja National Hospital, Mumbai
  - Gandhi Endocrinology & Diabetes Centre, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Deenanath Mangeshkar Hospital & Research Centre, Pune
  - Diabetes Care & Research Centre, Pune
  - Health & Research Centre, Trivendrum
  - Christian Medical College, Vellore